CLINICAL TRIAL: NCT07382453
Title: Effect of Poly（β-amino Ester）Hydrogel Loaded With tRNA-derived Fragments-antisense Oligonucleotides-exosomes on Patients With Diabetic Ocular Surface Diseases
Brief Title: Effect of PAE Hydrogel Loaded With tRF-ASO-Exo on Patients With Diabetic Ocular Surface Diseases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-L236
Record Dates: First submitted 2026-01-27; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Keratopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exo treatment (Experimental): Following a 14-day placebo run-in period-during which all subjects receive bilateral placebo eye drops (one drop per eye, twice daily, approximately 12 hours apart)-participants will receive active treatment for 84 days: Group 1 (Exo) receives 10 μg/drop of unmodified MSC-Exos.
  Interventions: Drug: Exosomes
- tRF-ASO-Exo treatment (Experimental): Following a 14-day placebo run-in period-during which all subjects receive bilateral placebo eye drops (one drop per eye, twice daily, approximately 12 hours apart)-participants will receive active treatment for 84 days:Group 2 (tRF-ASO-Exo) receives 10 μg/drop of tRF-ASO-engineered MSC-Exos.
  Interventions: Drug: tRNA-derived fragments-antisense oligonucleotides-exosomes
- tRF-ASO-Exo-PAE treatment (Experimental): Following a 14-day placebo run-in period-during which all subjects receive bilateral placebo eye drops (one drop per eye, twice daily, approximately 12 hours apart)-participants will receive active treatment for 84 days:Group 3 (tRF-ASO-Exo-PAE) receives 10 μg/drop of tRF-ASO-engineered MSC-Exos delivered via PAE hydrogel.
  Interventions: Drug: poly（β-amino ester）hydrogel loaded with tRNA-derived fragments-antisense oligonucleotides-exosomes

INTERVENTIONS:
Drug: Exosomes — Participants will receive artificial tears for 2 weeks to get the normalized baseline, followed by Exosomes 10ug/drop, two times a day for 84 days. The follow-up visit will be 12 weeks.
  Other Names: Exo
  Arms: Exo treatment
Drug: tRNA-derived fragments-antisense oligonucleotides-exosomes — Participants will receive artificial tears for 2 weeks to get the normalized baseline, followed by tRF-ASO-Exo 10ug/drop, two times a day for 84 days. The follow-up visit will be 12 weeks.
  Other Names: tRF-ASO-Exo
  Arms: tRF-ASO-Exo treatment
Drug: poly（β-amino ester）hydrogel loaded with tRNA-derived fragments-antisense oligonucleotides-exosomes — Participants will receive artificial tears for 2 weeks to get the normalized baseline, followed by tRF-ASO-Exo-PAE 10ug/drop, two times a day for 84 days. The follow-up visit will be 12 weeks.
  Other Names: tRF-ASO-Exo-PAE
  Arms: tRF-ASO-Exo-PAE treatment

SUMMARY:
The purpose of this study is to determine whether poly（β-amino ester）(PAE)hydrogel loaded with tRNA-derived fragments-antisense oligonucleotides-exosomes(tRF-ASO-Exo) could alleviate symptoms in patients with diabetic ocular surface diseases(DOSD).

DETAILED DESCRIPTION:
Diabetes mellitus is a highly prevalent, chronic systemic metabolic disorder affecting populations worldwide. According to the most recent data from the International Diabetes Federation (IDF), the global prevalence of diabetes among adults stands at 10.5%, whereas in China, it reaches 11.6%-corresponding to approximately 113.9 million affected adults, the highest absolute number globally. Diabetes-related systemic and ocular complications significantly impair patients' quality of life and impose substantial economic burdens on individuals, families, and healthcare systems, thereby constituting a pressing public health challenge requiring coordinated national and international action. Diabetic ocular surface disease (DOSD) represents one of the earliest and most frequently observed ocular complications of diabetes, often preceding other diabetic eye manifestations. Its incidence rises markedly with longer disease duration and suboptimal glycemic control. Notably, diabetic patients undergoing common ophthalmic procedures-including phacoemulsification for cataract, pterygium excision, and vitreoretinal surgery-are at heightened risk of postoperative keratoconjunctival disorders, which may progress to irreversible visual impairment or blindness, thereby threatening long-term ocular integrity. Among individuals with diabetes of ≥5 years' duration, over 60% develop moderate-to-severe dry eye or keratoconjunctival epithelial damage, clinically characterized by progressive symptoms including ocular dryness, foreign body sensation, photophobia, pain, and, in advanced cases, vision loss-collectively resulting in marked functional and quality-of-life deterioration.

Current clinical management of DOSD remains largely palliative, relying predominantly on artificial tear supplementation, secretagogues, and topical anti-inflammatory agents. However, these interventions do not address underlying neuroepithelial dysfunction and are limited by poor long-term adherence-reported rates fall below 50%-leading to suboptimal therapeutic outcomes. Consequently, the development of mechanism-targeted, disease-modifying therapies for DOSD is an urgent unmet clinical need.

Antisense oligonucleotides (ASOs) are synthetic, single-stranded RNA molecules designed to bind complementary tRNA-derived fragments (tRFs) with high specificity, thereby inhibiting their pathogenic activity. ASO-based therapeutics have demonstrated robust efficacy in neurodegenerative disorders, with several candidates having advanced to late-stage clinical trials. Engineered exosomes represent a next-generation drug delivery platform, offering enhanced nucleic acid loading capacity, improved pharmacokinetic stability, increased bioavailability, and superior tissue targeting compared with conventional exosomes or free small-molecule drugs. In ophthalmology, scalable production of engineered exosomes has opened new avenues for localized treatment of keratoconjunctival diseases. Furthermore, hydrogels provide physical encapsulation of nucleic acid therapeutics, shielding them from rapid enzymatic degradation in vivo; when combined with the intrinsic lipid bilayer of exosomes, this creates a synergistic "dual-barrier" protection system that markedly enhances therapeutic durability and clinical translatability. Poly(β-amino ester) (PAE) hydrogels-fabricated as biocompatible, three-dimensional scaffolds-retain the favorable properties of conventional hydrogels while additionally enabling sustained, controlled release, scalable manufacturing, and intrinsic neuroregenerative potential. In preclinical studies using a murine model of diabetic ocular surface disease, topical application of PAE hydrogel loaded with tRF-targeting ASO-engineered mesenchymal stem cell-derived exosomes (tRF-ASO-Exo) significantly attenuated ocular surface inflammation, promoted structural recovery of the corneal and conjunctival epithelium, and preserved corneal epithelial viability.

This study aims to evaluate a novel, non-invasive, topical hydrogel-based delivery system for tRF-ASO-loaded mesenchymal stem cell-derived exosomes (MSC-Exos) in patients with DOSD. The primary objective is to assess structural and functional ocular surface restoration using multimodal imaging and clinical metrics: anterior segment optical coherence tomography (AS-OCT), in vivo confocal microscopy (IVCM), slit-lamp-guided corneal fluorescein staining, and quantitative corneal sensitivity testing. Symptom improvement will be evaluated using the validated Ocular Surface Disease Index (OSDI). Secondary endpoints include tear secretion volume (Schirmer test), tear film breakup time (TBUT), ocular redness grading, tear meniscus height (via AS-OCT), and best-corrected visual acuity (BCVA).

A total of 30 participants will be enrolled and randomized into three intervention groups. Following a 14-day placebo run-in period-during which all subjects receive bilateral placebo eye drops (one drop per eye, twice daily, approximately 12 hours apart)-participants will receive active treatment for 84 days: Group 1 (Exo) receives 10 μg/drop of unmodified MSC-Exos; Group 2 (tRF-ASO-Exo) receives 10 μg/drop of MSC-Exos formulated in PAE hydrogel; and Group 3 (tRF-ASO-Exo-PAE) receives 10 μg/drop of tRF-ASO-engineered MSC-Exos delivered via PAE hydrogel-all administered twice daily. A 12-weeks follow-up will be conducted to monitor disease progression and durability of therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with fasting blood glucose ≥ 7.0 mmol/L or 2-hour postprandial blood glucose ≥ 11.1 mmol/L.

  2. Those who clearly understand and voluntarily participate in this study, and sign the written informed consent form themselves, and are able and willing to follow the instructions to participate in all trial evaluations and visits.

  3. Male subjects and female subjects of childbearing age must agree to use medically approved contraceptive measures during the trial and for 90 days after the trial. For female subjects who have not reached menopause or have been menopausal for less than two years, the pregnancy test must be negative.

  4. A history of severe dry eye symptoms (including one or more of the following subjective symptoms: dryness, foreign body sensation, burning sensation, fatigue, discomfort, redness, sudden eye pain, photophobia, tearing, blurred vision, and decreased corneal sensation) in both eyes for at least 180 days before the screening visit (Visit 0).

  5. Currently (within 30 days before Visit 0) using artificial tears to relieve dry eye-related symptoms, and artificial tears must be discontinued 72 hours before Visit 0.

  6. At Visit 0, the Chinese Dry Eye Questionnaire score is > 7 points or the total score of the Ocular Surface Disease Index is > 13 points.

  7. At Visit 0 and Visit 1, the dryness score is > 40 points. 8. At Visit 0, the best corrected visual acuity of both eyes is ≥ 4.3 (5-meter reading on the international standard logarithmic visual acuity chart, 5-point recording method).

  9. At Visit 0 and Visit 1, the corneal fluorescein staining score of at least one area of at least one eye is ≥ 2 points.

  10. At Visit 0 and Visit 1, the conjunctival redness score of at least one eye is ≥ 1 point.

  11. At the screening visit and baseline visit (Visit 0 and Visit 1), at least one eye of the same subject meets the following criteria: a. The corneal lower zone fluorescein staining score is ≥ 0.5 points; b. The Schirmer's test without anesthesia is ≥ 1 and ≤ 10 mm/5 min.

Exclusion Criteria:

1. Any past or current malignancy in or around the eye.
2. Dry eye traced to scarring (radiation, alkali burn, Stevens-Johnson, cicatricial pemphigoid) or goblet-cell loss (vitamin-A deficiency).
3. Active ocular allergy now or expected during the study.
4. Ocular or systemic infection at screening/baseline-fever, herpetic keratitis, or on antibiotics.
5. Prior immunodeficiency, HIV, hep B/C, active hep A, organ or bone-marrow transplant.
6. Any serious chronic illness the PI thinks could mess with endpoints-severe heart/lung disease, uncontrolled hypertension or diabetes.
7. Blood donation or major blood loss within 8 weeks of screening.
8. Active ocular rosacea, periorbital acne, or pterygium.
9. Lid problems-lagophthalmos, entropion, ectropion, or abnormal blink.
10. Clinically relevant slit-lamp findings needing treatment (conjunctivitis, trichiasis, conjunctivochalasis) that could skew results.
11. Eye surgery or laser (including YAG, meibomian thermopulsation, IPL) within 6 months of screening, or any such plan during the trial.
12. Punctal plugs (non-dissolvable within 90 days; dissolvable within 180 days) or planned plug procedures during the study.
13. Systemic steroids, immunomodulators, oral doxy/tetracycline within 90 days, or on-and-off use planned.
14. Topical glaucoma meds within 90 days.
15. Cyclosporine-A or lifitegrast drops within 42 days.
16. Drugs well known to dry the eye-diuretics, antidepressants, decongestants, antispasmodics, antihistamines, etc.-within 30 days or irregular use expected.
17. Active blepharitis/MGD therapy (lid scrubs, meibomian massage, warm compresses, systemic antibiotics) within 30 days or sporadic use planned.
18. Topical steroid or mast-cell stabilizer on the eye/face within 2 weeks.
19. Contact-lens wear within 7 days or intent to keep wearing them during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
corneal and conjunctival nerve density | 1day, 2 weeks, 6 weeks, 12 weeks
  In vivo confocal microscopy (IVCM) examination: All subjects underwent IVCM to assess corneal and conjunctival nerve density. Instruct the patient to fixate on a target, and the examiner slowly moves the objective lens until the vortex structure of the subbasal nerve plexus of the cornea can be seen.
Corneal sensitivity | 1day, 2 weeks, 6 weeks, 12 weeks
  Corneal sensitivity of the operated eye was evaluated by one examiner via a French Cochet-Bonnet aesthesiometer (Luneau Ophthalmologie), which consists of a calibrated nylon filament on a retractable shaft with a length scale. Longer filaments (lower bending force, weaker stimulus) indicate higher sensitivity. The sensitivity threshold was the maximum filament length evoking a reliable blink response. All tests were conducted in a standardized quiet indoor setting; patients kept eyes open with stable gaze during testing. Starting at 60 mm, the filament was perpendicularly applied to the central cornea, then shortened by 5 mm increments until consistent blinks occurred. Three measurements were taken, and corneal sensitivity was defined as the mean length of positive responses.
conjunctival goblet cell density | 1day, 2 weeks, 6 weeks, 12 weeks
  All participants underwent in vivo confocal microscopy (IVCM) assessment of conjunctival goblet cell density. Prior to imaging, subjects were instructed to maintain steady fixation on a standardized external target. The examiner systematically scanned the temporal bulbar conjunctiva approximately 3 mm from the corneal limbus, using the "section" scanning mode to acquire high-resolution images of the conjunctival epithelium-including the vortex region and its surrounding tissue within a 2-3 mm radius. To ensure optimal image quality and anatomical coverage, four non-overlapping image fields were captured per eye, each centered on a distinct location within a predefined small target zone. A sterile, single-use plastic cap was gently applied to the conjunctival surface prior to scanning to stabilize the ocular surface and minimize motion artifact. A total of 100-200 well-focused, artifact-free images were acquired for each examined eye.
Changes in Ocular Surface Staining | 1day, 2 weeks, 6 weeks, 12 weeks
  Ocular surface integrity was checked with a non-toxic dye at the slit lamp. Corneal and conjunctival staining were graded with the NEI photo atlas; lower scores mean less dry-eye damage. Change-from-baseline numbers were calculated for each eye, so a negative value equals improvement.
conjunctival vessel density and number of branches | 1day, 2 weeks, 6 weeks, 12 weeks
  AS-OCTA examination was performed to quantify conjunctival vasculature using anterior segment optical coherence tomography angiography. The anterior segment AS Angio 9×9 mm scan pattern with a resolution of 256×256 A-scans was selected for imaging and motion tracking. The scanning frame was positioned to intersect the corneal limbus, and the focal plane was adjusted until optimal visualization of the conjunctival layer was achieved. Superficial and deep conjunctival vascular plexuses were analyzed at depth ranges of 0-50 μm and 50-100 μm, respectively, with partial overlap between the two layers to account for transitional vascular networks. Vessel density and branching index were quantified using the device-integrated analytical software. Additionally, en face images were exported and further processed using ImageJ software (National Institutes of Health, USA) for supplementary image analysis.
Changes in Ocular Surface Disease Index (OSDI) Score | 1day, 2 weeks, 6 weeks, 12 weeks
  The Ocular Surface Disease Index (OSDI) is a validated 12-item questionnaire specifically designed to quantify the severity of dry eye symptoms in clinical settings. Its scoring range spans from 0 to 100, with lower scores correlating with a greater alleviation of dry eye-related discomfort. Baseline-adjusted OSDI scores were calculated, and a reduction of more than 10 points from the baseline value was defined as a clinically meaningful improvement in symptoms.

SECONDARY OUTCOMES:
Changes in tear secretion amount by Schirmer's Test | 1day, 2 weeks, 6 weeks, 12 weeks
  The examiner tucked a sterile paper strip beneath the lower lid, left it in place for the set time, then read the millimeters of strip the tears had traveled.
Changes in Tear break time | 1day, 2 weeks, 6 weeks, 12 weeks
  After a blink, the stopwatch ran until the first dry patch showed up on the ocular surface-time recorded in seconds.
Changes in best corrected visual acuity (BCVA) | 1day, 2 weeks, 6 weeks, 12 weeks
  to understand the effect of tRF-ASO-Exo-PAE on visual acuity
Changes in conjunctiva redness score | 1day, 2 weeks, 6 weeks, 12 weeks
  To explore the effect of tRF-ASO-Exo-PAE on conjunctiva. Under the slit lamp the investigator lined up each quadrant with the Allergan redness photos and handed out a 0-4 card: 0 = normal, vessels sharp; 1 = trace flush; 2 = mild; 3 = moderate; 4 = fiery severe-every step matched to its reference picture.

IPD SHARING:
Plan to Share IPD: No